CLINICAL TRIAL: NCT01668329
Title: Bio-clinical Evolutive Dynamic in Patients Suffering From Communitary Septic Shock (Biosepsis)
Acronym: BIOSEPSIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurDRC, Pr JF TIMSIT, University Hospital, Grenoble
Other Study IDs: 2009-A00822-55
Record Dates: First submitted 2010-07-08; First posted 2012-08-20 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2012-08

CONDITIONS: Immunocompetent Patient on Septic Shock
Keywords: Septic shock; Inflammatory process; Cytokines; Hormonal response; Oxydative stress
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — hormons, inflammatory markers, vitamines recovered from the patients serum.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Septic shock is a frequent pathology responsible for over 30000 deaths/year in France. Its outcome has not been improved despite the knowledge on inflammatory processes; a reason for these lack of results may lay on the lack of data on the precise dynamics of inflammatory and anti-inflammatory cascades and their consequences. We intend to achieve accurate monitoring of the inflammatory process on a small group of non-immunocompromised patients. Our goal is to obtain quality data, repeated over time, by limiting the technical variability.

DETAILED DESCRIPTION:
The aim is to obtain precise data on the dynamics of cytokines, oxydative stress and hormonal response on immunocompetent adults during septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years admitted in ICU.
* Clinical evidence of infection, suspected or proved, during the 48hrs following the hospital entry.
* Systemic inflammatory response syndrome.
* Shock defined as arterial hypotension (<90mmHg)not responding to adequated filling.

Exclusion Criteria:

* Minors
* Patient under guardianship or trusteeship
* Pregnant or lactating women
* Not affiliated to the social security
* Deprived of liberty by court decision
* Patients hospitalised without their approval
* Shock related to another cause than infection
* Long term corticothérapy
* On-going chemiothérapy, AIDS
* Bedridden patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All immunocompetent patients hospitalised in intensive care from the beginning of the septic shock state.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evolutive profile of the inflammatory response during septic shock | Hospitalisation in ICU

SECONDARY OUTCOMES:
Research for early prognosis factors | Hospitalisation in ICU

CONTACTS AND LOCATIONS:
Overall Officials: TIMSIT Jean FRANCOIS, PU/PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France